CLINICAL TRIAL: NCT04693650
Title: A Prospective, Multi-site, Randomized, Sham-Controlled, Double-Blind Trial With One-Way Crossover Designed to Assess the Effectiveness and Safety of the Gimer NeuroBlock SCS Trialing System for the Treatment of Chronic Back Pain and/or Lower Limb Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: GiMer Medical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: P20002
Record Dates: First submitted 2020-12-31; First posted 2021-01-05 (Actual); Last update posted 2023-02-27 (Actual); Status verified 2023-02

CONDITIONS: Chronic Pain; Low Back Pain; Lower Limb Pain
MeSH Terms: conditions — Chronic Pain; Low Back Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment group- UHF(+RF) stimulation (Experimental): Patients implanted with leads and be administered with UHF stimulation
  Interventions: Device: NeuroBlock UHF stimulation
- Control group (No Intervention): Patients implanted with lead receiving fake stimulation (no stimulation but same device procedure with test group)

INTERVENTIONS:
Device: NeuroBlock UHF stimulation — NeuroBlock ultrahigh frequency (UHF) stimulation with 500kHz intra-pulse
  Other Names: +RF (plus RF, pulsed RF)
  Arms: Treatment group- UHF(+RF) stimulation

SUMMARY:
This study is a prospective, multi-site, randomized, shamcontrolled, double-blind trial with one-way crossover designed to assess the effectiveness and safety of the Gimer NeuroBlock SCS Trialing System for the treatment of chronic back pain and/or lower limb pain. The NeuroBlock SCS Trialing System is an ultra-high frequency SCS device for the treatment of patients with chronic back pain and/or lower limb pain who are refractory to conservative pain management. After screening procedures, eligible subjects will enter the study which is comprised of a 1-week randomized testing period, a 1-week follow-up period and 2-week observation period.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 20
2. Subject has been diagnosed with chronic, intractable pain of the trunk and/or limb(s) and is refractory to conservative therapy for a minimum of six months prior to the screening/baseline visit.
3. Subject has an average pain score of back or leg ≥ 5 or maximum pain score of back or leg ≥ 7 on the Visual Analogue Scale (VAS).
4. Subject is willing and able to comply with the procedure and requirements of this trial.
5. The subject is able to understand and provide informed consent, and has signed their written informed consent in accordance with IRB requirements.

Exclusion Criteria:

1. Subject has the following conditions by investigator's discretion at screening visit or during the last 3 months:

   1. has the mental or psychological condition that affects pain perception or
   2. has difficulty performing objective pain assessment or lack of suitability for participation in the study.
2. Subject has exhibited unstable pain condition within the past 28 days as interviewed by Investigator.
3. Subject has a currently diagnosed coagulation disorder, bleeding diathesis, progressive peripheral vascular disease with PLT < 100,000/μl or INR > 1.4 at screening visit.
4. Subject has unstable pain medication(s) for at least 28 days at investigator's discretion.
5. Subject currently has an active implantable device including ICD, pacemaker, spinal cord stimulator or intrathecal drug pump or subject requires magnetic resonance imaging (MRIs) or diathermy.
6. Subject has a current diagnosis of cancer with active symptoms.
7. Subject has a known terminal illness with life expectancy less than one year.
8. Subject has a systematic or local infection, which may increase study risk.
9. Subject currently has an indwelling device that may pose an increased risk of infection.
10. Subject is pregnant or breast feeding.
11. Subject has a medical history of drug or alcohol addiction within the past 2 years.
12. Subject has participation in any investigational study in the last 30 days or current enrollment in any trial.
13. Subject is currently involved in an injury claim law suit or medically related litigation, including workers compensation.
14. Subject is a prisoner.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2022-02-01 (Actual); Study Completion 2022-04-01 (Actual)

PRIMARY OUTCOMES:
Effectiveness: Responder Rate | 2 weeks
  The responder rate of the test group and control group at the 2-week visit
Safety: AEs and SAEs | 4 weeks
  Incidence of adverse events (AEs) and serious AEs (SAEs)

CONTACTS AND LOCATIONS:
Locations (4):
- Taiwan (4):
  - China Medical University Hospital, Taichung
  - Mackay Memorial Hospital, Taipei
  - National Taiwan University Hospital, Taipei
  - Veterans General Hospital-Taipei, Taipei